CLINICAL TRIAL: NCT03324243
Title: A Phase II Study of Crenolanib With Fludarabine and Cytarabine in Pediatric Patients With Relapsed/Refractory FLT3-Mutated Acute Myeloid Leukemia
Brief Title: A Study of Crenolanib With Fludarabine and Cytarabine in Pediatric Patients With Relapsed/Refractory FLT3-Mutated Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn: Study halted prior to enrollment of first participant
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARO-014
Record Dates: First submitted 2017-10-18; First posted 2017-10-27 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Relapsed/Refractory FLT3-mutated AML
MeSH Terms: conditions — Recurrence | interventions — crenolanib; fludarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crenolanib (Experimental)
  Interventions: Drug: Crenolanib; Drug: Fludarabine; Drug: Cytarabine

INTERVENTIONS:
Drug: Crenolanib — 66.7 mg/m2 three times a day (TID)
  Other Names: Crenolanib besylate
Drug: Fludarabine — 30 mg/m2/day, intravenous infusions over 30 mins.
Drug: Cytarabine — 2000 mg/m2/day, intravenous infusions over 1-3 hours.

SUMMARY:
This is a phase II, multicenter, single-arm study to assess the safety and feasibility of combining crenolanib with fludarabine and cytarabine chemotherapy in pediatric patients with relapsed/refractory FLT3-mutated AML. Patients will receive up to two courses of salvage chemotherapy with fludarabine, cytarabine, and crenolanib. Response will be assessed between day 29-43 of each course.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 1 years and ≤ 21 years
2. Confirmed diagnosis of AML according to World Health Organization (WHO) 2016 classification
3. Definitive evidence of a FLT3-ITD and/or FLT3-TKD (D835/I836) mutation at the time of enrollment
4. Patients must have histologically or molecularly confirmed relapsed or refractory AML
5. Karnofsky or Lansky performance score ≥ 50. Use Karnofsky for patients > 16 years old and Lansky for patients ≤ 16 years of age.
6. Adequate renal function, defined as:

   * Creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73 m2 or
   * Normal serum creatinine based on age/gender
7. Adequate liver function, defined as:

   * Serum total bilirubin ≤ 1.5x ULN for age,
   * Serum aspartate aminotransferase (AST) ≤ 3.0x ULN for age, and
   * Serum alanine aminotransferase (ALT) ≤ 3.0x ULN for age.

Exclusion Criteria:

1. Patients with any of the following current or previous diagnoses:

   * Acute promyelocytic leukemia (APL)
   * Down syndrome
   * DNA fragility or bone marrow failure syndromes (such as Fanconi anemia, Bloom syndrome, Kostmann syndrome, or Shwachman syndrome)
   * AML secondary to prior MDS/MPN, including chronic myelomonocytic leukemia and juvenile myelomonocytic leukemia
   * Blastic plasmacytoid dendritic cell neoplasm
   * Acute leukemia of ambiguous lineage
   * B-lymphoblastic leukemia/lymphoma
   * T-lymphoblastic leukemia/lymphoma, including early T-cell precursor lymphoblastic leukemia (ETP-ALL)
2. Patients who are refractory to first line (induction and re-induction) and a second line (1st salvage) treatment for AML.
3. Patients who have received more than 1 prior allogeneic HSCT
4. Patients will be excluded if they have a systemic fungal, bacterial, viral or other infection of which they exhibit ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment.
5. Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
6. Known severe liver disease (e.g. cirrhosis, non-alcoholic steatohepatitis, sclerosing cholangitis or hyperbilirubinemia)
7. Known, active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
8. Currently receiving prophylactic treatment of hepatitis B with anti-viral therapy
9. Known infection with human immunodeficiency virus (HIV)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing ≥ Grade 3 adverse events as assessed by CTCAE v4.0 | From study entry to 30 days post-treatment
Number of patients experiencing Grade 4 adverse events related to crenolanib as assessed by CTCAE v4.0 | 60 days
Rate of early mortality | 60 days
  Number of patients who died within 60 days of start of therapy

SECONDARY OUTCOMES:
Event-free survival (EFS) | 4 years
  EFS is defined as the time from the date of start of treatment to the date of failure to achieve a remission, relapse, or death from any cause.
Relapse-free survival (RFS) | 4 years
  RFS is defined as the time from the date of remission to date of relapse or death.
Overall survival (OS) | 4 years
  OS is defined as the time from the date of start of treatment until death.

IPD SHARING:
Plan to Share IPD: No